CLINICAL TRIAL: NCT06401356
Title: An Open-Label, Multicenter, Extension Study for Patients Previously Enrolled in Studies With Pelabresib
Brief Title: An Extension Study for Patients Previously Enrolled in Studies With Pelabresib
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDAK539A12001B; CNST0610C210 (Other: Constellation Pharmaceuticals); 2023-508950-24-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Hematologic Malignancy; Solid Tumor; Advanced Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — CPI-0610

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pelabresib (Experimental): All eligible participants will receive continued treatment with pelabresib as administered in the relevant parent study.
  Participants previously enrolled in studies with pelabresib who discontinued treatment with placebo or pelabresib may be enrolled in this extension study for the purpose of survival follow-up.
  Interventions: Drug: Pelabresib

INTERVENTIONS:
Drug: Pelabresib — Small molecule inhibitor of bromodomain and extraterminal (BET) protein
  Other Names: CPI-0610

SUMMARY:
The purpose of this study is to evaluate the long-term safety and the clinical benefit of pelabresib in patients with hematological and/or solid tumor indications or advanced malignancies. Additionally, participants previously enrolled in studies with pelabresib who received placebo or participants who discontinued pelabresib (for any other reason than participating in this extension study), may be enrolled in this extension study to evaluate the survival and leukemia-free survival (for patients with hematological malignancies) or only the Survival Follow-up (for all the other patients).

DETAILED DESCRIPTION:
The study will collect and monitor ongoing efficacy information with regard to disease and survival status, as well as safety information with regard to AEs, including SAEs and AEs of special interest (AESI).

Patients are eligible to continue pelabresib treatment as long as the regimen is tolerated, and the patient does not meet any of the discontinuation criteria.

There will be an eligibility check period of up to 28 days for this extension study. Patients who fulfill the inclusion and exclusion criteria are eligible for the study. After the patient willingly provides consent, eligibility will be assessed by the investigator and treatment with pelabresib can be started at the same dose and dosing schedule that was applied in the parent study in the last cycle prior to EOT unless there is need for dose adjustment due to toxicity.

A patient is considered to have completed the study after completion of all visits as defined in the Schedule of Assessments (SoA) as per protocol, including the Safety Follow-up visit and Survival Follow-up.

The Safety Follow-up period is the interval between the EOT visit and the scheduled Safety Follow-up visit, which should occur 30 days (±3 days) after the last dose of pelabresib. For patients who switch from investigational pelabresib to commercial pelabresib treatment, the Safety Follow-up period is the time from the last dose of investigational pelabresib until the first dose of commercial pelabresib. The treatment start date with commercial pelabresib will be considered the date of "early Safety Follow-up termination." All patients will be followed for AEs and SAEs for 30 days (±3 days) following the last dose of pelabresib on the extension study or until the initiation of a new anticancer therapy, whichever occurs first.

Reasonable efforts should be made to have the patient return for the Safety Follow-up visit and review any AEs that may occur during this period. If the patient cannot return to the site for the Safety Follow-up visit, then the patient should be contacted by telephone for assessment of AEs.

The end of study will occur when all parent studies have been closed with no further patients expected to be enrolled into the extension study, and the last patient in the extension study has permanently discontinued study treatment (investigational pelabresib) and has completed the Safety Follow-up visit or is designated as lost to follow-up, died, or has withdrawn consent, whichever comes first. The sponsor reserves the right to close a study site or terminate the study at any time for any reason at the sole discretion of the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Eligibility for Ongoing Pelabresib Treatment

   * Able to provide signed informed consent, agreeing to all protocol and ICF requirements.
   * At least 18 years old and legally able to consent in the study's jurisdiction.
   * Previously enrolled and currently receiving pelabresib in a parent study.
   * Demonstrating clinical benefit from pelabresib, as judged by the investigator.
   * Willing and able to follow all study visits, treatments, and procedures.
   * Agree to avoid pregnancy or fathering children:

     * Men: Must use highly effective contraception (≥99% effective) and avoid sperm donation from eligibility check through 94 days post-treatment.
     * Women of childbearing potential (WOCBP): Must test negative for pregnancy at eligibility, use highly effective contraception through 184 days post-treatment, undergo regular pregnancy testing, and avoid breastfeeding and oocyte donation during this period.
     * Women not of childbearing potential (surgically sterile or postmenopausal ≥12 months without other cause) are eligible.

   Note: Women with amenorrhea due to chemo/radiotherapy are considered WOCBP and must use contraception.
2. Eligibility for Survival Follow-up

   * Provide signed informed consent, agreeing to all protocol and ICF requirements.
   * Are at least 18 years old and legally able to consent.
   * Were previously enrolled in a pelabresib clinical study.
   * Are willing and able to comply with follow-up procedures.

Exclusion Criteria:

1. Eligibility for Ongoing Pelabresib Treatment

   * Legally institutionalized or under judicial protection.
   * Enrolled in another interventional clinical trial (excluding the parent study).
   * History of hypersensitivity to pelabresib, its excipients, or similar drugs.
   * Significant gastrointestinal issues (e.g., active IBD, unresolved nausea/vomiting/diarrhea > Grade 1) that may affect drug absorption.
   * Any medical condition deemed unsuitable by the investigator.
   * Uncontrolled illness or condition that may compromise safety or protocol compliance.
   * Received systemic anticancer or investigational treatment (excluding parent study drug or hormonal therapy) within 2 weeks or 5 half-lives before first dose. (Hydroxyurea/anagrelide allowed up to 24 hours prior.)
   * Received hematopoietic growth factors or androgenic steroids within 4 weeks before first dose.
   * Used strong CYP3A4 inhibitors/inducers (e.g., St. John's wort) within 2 weeks before first dose. Use during treatment is prohibited.
   * Female participants who are pregnant, breastfeeding, or not using required contraception.
   * Male participants who do not agree to use contraception or refrain from sperm donation as specified.
   * Unwilling or unable to comply with the study protocol.
2. Eligibility for Survival Follow-up • They are legally institutionalized or under judicial protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2027-06-02 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) and serious TEAEs | 5 years
  To evaluate long-term safety in patients who are receiving pelabresib
Survival Follow-up | 5 years
  Survival Follow-up consists of Survival and Leukemia-Free Survival Follow-up. All participants in the extension study will be followed up for Survival, while participants with hematological malignancies will be followed up for Survival and Leukemia-Free Survival. In addition, participants who will not receive pelabresib treatment may enter this extension protocol to be only followed up for Survival.
Duration of Response (DoR) | 5 years
  DOR defined as the time from the date of first response to the date of confirmed disease progression
Progression-free survival (PFS) | 5 years
  PFS defined as the time from first dose to confirmed disease progression or death, whichever occurs first.
Leukemia-free survival (LFS) | 5 years
  LFS defined as the time from first dose to the date of leukemic transformation or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- United States (6):
  - Hematologic Malignancy/Stem (Department of Medicine, Division of Hematology/Oncology), Los Angeles, California
  - Mayo Clinic (Cancer Clinical Research Office), Jacksonville, Florida
  - Northwestern Memorial Hospital (Oncology), Chicago, Illinois
  - UMHS - University of Michigan Medical Center (Radiation Oncology), Ann Arbor, Michigan
  - Mount Sinai Hospital - Oncology, New York, New York
  - Weill Cornell Medicine - New York Presbyterian Hospital (Oncology), New York, New York
- Belgium (2):
  - ZNA Cadix-Hematology, Antwerp
  - Az St-Jan Brugge-Oostende A.V., Bruges
- Italy (3):
  - AOU Careggi (Department of Experimental and Clinical Medicine), Florence
  - Azienda Ospedaliero - Universitaria Maggiore della Carità (SCDU Ematologia), Novara
  - AO Ospedale di Circolo, PO Varese (Ematologia), Varese
- Amsterdam UMC location Vumc (Hematology), Amsterdam, Netherlands
- United Kingdom (3):
  - Cardiff and Vale University Health Board - University Hospital Wales (Hematology), Cardiff
  - Beatson West of Scotland Cancer Centre (Hematology), Glasgow
  - Guys and St Thomas' Hospital - Haematology, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com